CLINICAL TRIAL: NCT07062926
Title: Comparative Effects of Spencer Muscle Energy Technique Versus Post Facilitation Stretch on Pain, Range of Motion, and Functional Disability Among Fast Bowlers With Shoulder Pain
Brief Title: Comparative Effects of Spencer Muscle Energy Technique Versus Post Facilitation Stretch Among Fast Bowlers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0447
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Sports Physical Therapy
Keywords: spencer technique, post facilitation stretch, shoulder pain.
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Intervention Model Description: Randomized control design
Who Masked: Participant
Masking Description: The participants are blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spencer Muscle Energy Technique (Experimental): 16 participants will undergo spencer muscle energy technique three times a week over a four-week period.Various movement patterns will performed, and the treatment duration will be 30 minutes.
  Interventions: Other: Spencer Muscle Energy Technique
- Post Facilitation Stretch (Experimental): 16 participants will undergo Post facilitation stretching process was repeated 5 times with 10 second interval between each stretch. The whole treatment session was around 20 minute.
  Interventions: Other: Post Facilitation Stretch

INTERVENTIONS:
Other: Spencer Muscle Energy Technique — Spencer muscle energy technique participants will receive a hot pack for 7-10 minutes followed by their respective treatments, three times a week for four weeks. Group A will undergo Spencer Muscle Energy Technique for 30 minutes
  Other Names: Assigned
  Arms: Spencer Muscle Energy Technique
Other: Post Facilitation Stretch — Post facilitation stretch participants will receive a hot pack for 7-10 minutes followed by their respective treatments, three times a week for four weeks.post facilitation stretching process was repeated 5 times with 10 second interval between each stretch.
  Other Names: Assigned
  Arms: Post Facilitation Stretch

SUMMARY:
This study compares the effectiveness of Spencer Muscle Energy Technique and Post Facilitation Stretch in reducing shoulder pain in 32 fast bowlers aged 18-35. Participants will receive treatment three times a week for four weeks. Pain, shoulder mobility, and functional ability will be measured before and after the intervention to identify the more effective technique

DETAILED DESCRIPTION:
This randomized clinical trial aims to compare the effectiveness of the Spencer Muscle Energy Technique and Post Facilitation Stretch in treating shoulder pain among fast bowlers. A total of 32 fast bowlers aged 18-35 years with chronic shoulder pain will be recruited from the Pakistan Sports Board, Lahore. Participants will be randomly divided into two groups, each receiving one of the two treatments three times a week for four weeks, preceded by hot pack application. Pain, shoulder range of motion, and functional disability will be assessed before and after the intervention using the Visual Analogue Scale, inclinometer, and Quick-DASH questionnaire. The study seeks to determine which technique offers better outcomes for managing shoulder pain in fast bowlers.

ELIGIBILITY:
Inclusion Criteria:

* Fast bowlers

  * Both male and female.
  * aged 18-35 years.
  * Stiff painful shoulder joint for at least 3 months.
  * Willingness to participate in the study and provide informed consent.

Exclusion Criteria:

* ● Rotator cuff tears.

  * Rheumatoid and gouty arthritis.
  * Tumors of the shoulder region.
  * Reflex sympathetic dystrophy of the shoulder.
  * Thoracic outlet syndrome, peripheral nerve injuries, shoulder girdle fractures, dislocations.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-06-25 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | 4 Weeks
  Pain intensity was measured using a 10-cm VAS, where 0 indicates "no pain" and 10 indicates "worst imaginable pain." Scores were recorded at baseline and after 4 weeks of intervention.
Range of Motion | 4 Weeks
  Active shoulder flexion, abduction, and external rotation were assessed using a digital inclinometer. Each movement was measured three times and averaged. Assessments were conducted at baseline and after the intervention period.
Quick Disabilities of the Arm, Shoulder and Hand (Quick-DASH) Score | 4 Weeks
  A validated questionnaire used to assess functional disability of the upper limb. It consists of 11 items scored on a 5-point Likert scale. Final scores range from 0 (no disability) to 100 (most severe disability). It was recorded pre- and post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Syeda Tehreem Fatima, DPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghisi D, Boschetto G, Spinelli AM, Giannone S, Frugiuele J, Ciccarello M, Bonarelli S. Spinal anaesthesia with Chloroprocaine HCl 1% for elective lower limb procedures of short duration: a prospective, randomised, observer-blind study in adult patients. BMC Anesthesiol. 2021 Feb 20;21(1):58. doi: 10.1186/s12871-021-01279-9. PMID 33610175
- [Background] Kawabata Y, Ikegami H. Genetics of fulminant type 1 diabetes. Diabetol Int. 2020 Sep 21;11(4):315-322. doi: 10.1007/s13340-020-00468-0. eCollection 2020 Oct. PMID 33088637
- [Background] Su PY, Su WW, Hsu YC, Wang SY, Chiu PF, Yen HH. Micro-Elimination of Hepatitis C among Patients with Kidney Disease by Using Electronic Reminder System-A Hospital-Based Experience. J Clin Med. 2022 Jan 14;11(2):423. doi: 10.3390/jcm11020423. PMID 35054120
- [Background] Chia M. PRIDE for PLAY: Personal Responsibility in Daily Effort for Participation in Lifelong Activity for Youths. A Singaporean Context. J Sports Sci Med. 2007 Sep 1;6(3):374-9. PMID 24149424
- [Background] Phansopkar P, Qureshi MI. Impact of Spencer Technique on Pain, Range of Motion, and Functional Disability in Patients With Frozen Shoulder: A Pilot Study. Cureus. 2024 Jan 30;16(1):e53263. doi: 10.7759/cureus.53263. eCollection 2024 Jan. PMID 38435910
- [Background] Iqbal M, Riaz H, Ghous M, Masood K. Comparison of Spencer muscle energy technique and Passive stretching in adhesive capsulitis: A single blind randomized control trial. J Pak Med Assoc. 2020 Dec;70(12(A)):2113-2118. doi: 10.5455/JPMA.23971. PMID 33475581